CLINICAL TRIAL: NCT00436566
Title: Phase II Study of Cardiac Safety and Tolerability of an Adjuvant Chemotherapy Plus Trastuzumab With Lapatinib in Patients With Resected HER2 + Breast Cancer
Brief Title: Doxorubicin and Cyclophosphamide Followed By Trastuzumab, Paclitaxel, and Lapatinib in Treating Patients With Early-Stage HER2-Positive Breast Cancer That Has Been Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: CDR0000533793; P30CA015083 (NIH); RC0639 (Other: Mayo Clinic Cancer Center); 06-004049 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Results first posted 2012-11-21 (Estimated); Last update posted 2022-08-05 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer; Cardiac Toxicity
Keywords: cardiac toxicity; male breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity; Breast Neoplasms, Male | interventions — Trastuzumab; Cyclophosphamide; Doxorubicin; Lapatinib; Paclitaxel; Gene Expression Profiling; Reverse Transcriptase Polymerase Chain Reaction; Fluorophotometry; Mass Spectrometry; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: trastuzumab
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: lapatinib ditosylate
Drug: paclitaxel
Genetic: gene expression analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: fluorophotometry
Other: laboratory biomarker analysis
Other: mass spectrometry
Procedure: adjuvant therapy
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin, cyclophosphamide, and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving combination chemotherapy together with trastuzumab and lapatinib after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This randomized phase II trial is studying the side effects and how well giving doxorubicin together with cyclophosphamide followed by trastuzumab, paclitaxel, and lapatinib works in treating patients with early-stage HER2-positive breast cancer that has been removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the cardiac safety of adjuvant therapy comprising doxorubicin hydrochloride and cyclophosphamide followed by paclitaxel, trastuzumab (Herceptin®), and lapatinib ditosylate in patients with resected early-stage HER2-positive breast cancer.

Secondary

* Determine the adverse event profile of this regimen in these patients.
* Determine the cumulative incidence of cardiac events in patients treated with this regimen.
* Determine the LVEF in patients treated with this regimen.
* Determine the disease-free and overall survival of patients treated with this regimen.
* Compare selected quality-of-life (QOL) questionnaires in these patients.
* Evaluate QOL of patients treated with this regimen.
* Determine the cumulative incidence of pulmonary events in patients treated with this regimen.

Tertiary

* Compare Veridex CellSearch system vs quantitative reverse transcriptase polymerase chain reaction for detecting circulating tumor cells.
* Determine the relationship between serum levels of HER1 and HER2 and response to treatment.
* Evaluate cardiac markers (i.e., troponin-T, troponin-I, brain natriuretic peptide, and creatine kinase MB isoenzyme) at baseline.
* Determine the association between abnormal levels of cardiac markers and incidence of cardiac adverse events.
* Evaluate patterns of 500 metabolites in plasma in patients treated with this regimen and determine the association between metabolite patterns/molecular signatures and cardiotoxicity.
* Determine the time course of these molecular signatures and evaluate whether they are accurate predictors of cardiotoxicity that precede other evidence of cardiotoxicity (e.g., changes in left ventricular function seen by echocardiogram or MUGA scan).
* Compare metabolic signatures of cardiotoxicity with known laboratory evidence of cardiac damage (e.g., troponins or brain natriuretic peptide) in terms of sensitivity and specificity.

OUTLINE: This is a randomized, pilot, multicenter study. Patients are stratified according to educational level (less than high school vs high school or GED vs formal education beyond high school).

Patients receive doxorubicin hydrochloride IV and cyclophosphamide IV on day 1. Treatment repeats every 2-3 weeks for 4 courses. Patients then receive paclitaxel IV over 60 minutes and trastuzumab (Herceptin®) IV over 90 minutes on days 1, 8, and 15 and oral lapatinib ditosylate on days 1-21. Treatment with paclitaxel, trastuzumab, and lapatinib repeats every 3 weeks for up to 4 courses. Patients then receive trastuzumab IV over 30-90 minutes on day 1 and oral lapatinib ditosylate on days 1-21. Treatment with trastuzumab and lapatinib ditosylate repeats every 3 weeks for up to 12 courses.

Patients complete Linear Anologue Self Assessment (LASA) and Symptoms Distress Scale (SDS) questionnaires, including fatigue, diarrhea, and rash assessment, at baseline, after 2-3, 5-6, and 18 months of treatment, and 5 years after completion of treatment. Patients are also randomized to 1 of 2 arms to complete additional quality of life questionnaires at these same time points.

* Arm I: Patients complete EORTC QLQ-C30 and EORTC QLQ-BR23 questionnaires.
* Arm II: Patients complete FACT-B questionnaire. Blood samples are acquired periodically throughout and at the completion of study treatment. Samples are analyzed for circulating tumor cells by Veridex CellSearch system, quantitative reverse transcriptase polymerase chain reaction, and liquid chromatography with tandem mass spectrometry, soluble HER1- and HER2-receptor concentrations, circulating cardiac markers, and metabolic markers for possible correlation with cardiac events.

After completion of study treatment, patients are followed periodically for up to 10 years.

PROJECTED ACCRUAL: A total of 109 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of early-stage breast cancer

  * HER2 positive by immunohistochemistry (IHC) (3+) or fluorescent in situ hybridization (FISH)

    * Ductal carcinoma in situ (DCIS) components should not be counted in the determination of degree of IHC staining or FISH amplification
* No locally advanced tumors (i.e., T4) at diagnosis, including the following:

  * Tumors fixed to chest wall
  * Peau d'orange
  * Skin ulcerations or nodules
  * Clinical inflammatory changes (e.g., diffuse brawny cutaneous induration with an erysipeloid edge)
* Has undergone mastectomy or lumpectomy with axillary node or sentinel node dissection within the past 84 days

  * Patients who have undergone a mastectomy must meet the following criteria:

    * No evidence of gross or microscopic tumor (i.e., invasive DCIS) at the surgical resection margins noted in final surgery or pathology reports

      * Patients with close margins are eligible
    * Radiation therapy is required for 4 or more positive lymph nodes and must be started after completion of chemotherapy
  * Patients who have undergone a lumpectomy with axillary node or sentinel node dissection must meet the following criteria:

    * No evidence of invasive cancer or DCIS at the surgical resection margins
    * No gross residual adenopathy
    * Planning to undergo radiation therapy to the breast with or without regional lymphatics after completion of chemotherapy
* No active hepatic or biliary disease

  * Patients with liver metastases, stable chronic liver disease, Gilbert's syndrome, or asymptomatic gallstones are eligible
* Hormone receptor status:

  * Estrogen receptor and progesterone receptor status known

PATIENT CHARACTERISTICS:

* Male or female
* Menopausal status not specified
* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10.0 g/dL
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* LVEF ≥ 50% by MUGA scan or echocardiogram
* Able to complete questionnaire(s) by themselves or with assistance
* Able and willing to provide blood and tissue samples
* No known sensitivity to benzyl alcohol
* No sensory neuropathy ≥ grade 2
* No active cardiac disease, including any of the following:

  * Myocardial infarction within the past 6 months
  * Prior or concurrent congestive heart failure
  * Prior or concurrent arrhythmia or cardiac valvular disease requiring medications or that is clinically significant
  * Uncontrolled hypertension, defined as diastolic blood pressure (BP) >100 mm Hg or systolic BP > 200 mm Hg on 2 separate occasions ≥ 14 days apart
  * Clinically significant pericardial effusion
  * Prior or concurrent uncontrolled or symptomatic angina
  * Other cardiac condition that, in the opinion of the treating physician, would put the patient at hazardous risk
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition as lapatinib ditosylate
* No uncontrolled intercurrent illness including, but not limited to, the following:

  * Ongoing or active infection
  * Psychiatric illness or social situations that would preclude study compliance
* Able to swallow and retain oral medication

  * No history of gastrointestinal (GI) disease resulting in an inability to take oral medication, including any of the following:

    * Malabsorption syndrome
    * Requirement for IV alimentation
    * Prior surgical procedures affecting absorption
    * Uncontrolled inflammatory GI disease (e.g., Crohn's disease or ulcerative colitis)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy, radiation therapy, immunotherapy, or biotherapy for breast cancer
* No primary breast radiation therapy as part of breast-conserving treatment
* No prior anthracycline or taxane therapy for any malignancy
* No prior epidermal growth factor receptor-targeting therapies (e.g., gefitinib, cetuximab, erlotinib hydrochloride, rituximab, trastuzumab [Herceptin®], lapatinib ditosylate, panitumumab, or nimotuzumab)
* At least 14 days since prior and no concurrent CYP3A4 inducers, including the following:

  * Rifamycin-class antibiotics (e.g., rifampin, rifabutin, or rifapentine)
  * Anticonvulsants (e.g., phenytoin, carbamazepine, or barbiturates [e.g., phenobarbital])
  * Antiretrovirals (e.g., efavirenz or nevirapine)
  * Glucocorticoids (e.g., oral cortisone, hydrocortisone, prednisone, methylprednisolone, or dexamethasone)

    * Daily oral dexamethasone ≤ 1.5 mg (or equivalent) allowed
  * Modafinil
  * Hypericum perforatum (St. John's wort)
* At least 7 days since prior and no concurrent CYP3A4 inhibitors, including the following:

  * Antibiotics (e.g., clarithromycin, erythromycin, or troleandomycin)
  * Antifungals (e.g., itraconazole, ketoconazole, fluconazole [> 150 mg daily], or voriconazole)
  * Antiretrovirals and protease inhibitors (e.g., delaviridine, nelfinavir, amprenavir, ritonavir, indinavir, saquinavir, or lopinavir)
  * Calcium channel blockers (e.g., verapamil or diltiazem)
  * Antidepressants (e.g., nefazodone or fluvoxamine)
  * Gastrointestinal agents (e.g., cimetidine or aprepitant)
  * Grapefruit and grapefruit juice
* At least 6 months since prior and no concurrent amiodarone
* No herbal or alternative medicines or supplements ≥ 14 days before, during, and for 30 days after completion of study treatment
* No concurrent hormonal agents (e.g., birth control pills, ovarian hormonal replacement therapy, or raloxifene)

  * Adjuvant hormonal agents (e.g., tamoxifen, aromatase inhibitors) allowed after completion of chemotherapy as part of treatment for breast cancer
* No concurrent antiretroviral therapy for HIV-positive patients
* No concurrent digitalis or beta-blockers for congestive heart failure
* No concurrent arrhythmia or angina pectoris medication
* No other concurrent investigational agents or anticancer therapies, including cytotoxic agents or immunotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2007-03-16 (Actual); Primary Completion 2009-04 (Actual); Study Completion 2019-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edith A. Perez, MD, Study Chair — Mayo Clinic; Donald W. Northfeld, MD, Principal Investigator — Mayo Clinic; James N. Ingle, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic Cancer Research Consortium, Rochester, Minnesota, United States

REFERENCES:
- [Result] McCullough A, Dueck A, Chen B, et al.: HER-2 central confirmatory testing using ASCO/CAP guidelines for trastuzumab/lapatinib trial MCCR RC0639. [Abstract] J Clin Oncol 27 (Suppl 15): A-e11527, 2009.
- [Result] Palmieri FM, Dueck AC, Johnson DB, et al.: Cardiac safety of lapatinib given concurrently with paclitaxel and trastuzumab as part of adjuvant therapy for patients with HER2+ breast cancer: Pilot data from the Mayo Clinic Cancer Research Consortium Trial RC0639. [Abstract] 32nd Annual San Antonio Breast Cancer Symposium, December 9-13, 2009, San Antonio, Texas. A-3086, 2009.
- [Result] Johnson BS, Dueck AC, Dakhil SR, et al.: Tolerability of lapatinib given concurrently with paclitaxel and trastuzumab as part of adjuvant therapy in patients with resected HER2+ breast cancer: initial safety data from the Mayo Clinic Cancer Research Consortium trial RC0639. [Abstract] 31st Annual San Antonio Breast Cancer Symposium, December 10-14, 2008, San Antonio, Texas. A-2109, 2008.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One-hundred and twenty-two (122) participants were recruited between April 2007 and October 2008 at Mayo Clinic. Ten (10) participants were deemed ineligible due to HER-2+ not corroborated by the central laboratory evaluation. These 10 participants and 3 participants (those who did not completed the treatment) were excluded from all analysis.
Groups:
- AC/PTL: Standard doxorubicin and cyclophosphamide (AC) followed by weekly paclitaxel (80 mg/m^2) x 12 with concurrent standard dose trastuzumab (weekly x 12, then repeat 3 weeks for an additional 9 months) plus daily lapatinib (modified to 750 mg during Paclitaxel + Trastuzumab + Lapatinib (PTL) and 1000 mg during trastuzumab + lapatinib (TL)) for a total of 12 months.
Period: Overall Study
Arm/Group | AC/PTL
Started | 112
Completed | 109
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | AC/PTL
Number analyzed (Participants) | 109
Age, Continuous [Median (Full Range); unit: years] | 51 [28 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 94
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 109
Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: participants] — Performance Status Grade:
  0=Fully active, able to carry on all predisease activities without restriction (Karnofsky 90-100); 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work (Karnofsky 70-80).
  participants
    0 | 91
    1 | 18
T Stage [Number; unit: participants]
  T1=Tumor <=2 cm (3/4 of an inch) across | 43
  T2=2cm < Tumor <5 cm across | 58
  T3=Tumor > 5 cm across | 6
  Missing | 2
Nodal Status [Number; unit: participants] — N0=Node negative (either by negative sentinel node or by axillary dissection); N1=Node positive (axillary nodal dissection with 1-3 + nodes); N2=Node positive (axillary nodal dissection with 4-9 + nodes); N3=Node positive (axillary nodal dissection with 10+ nodes); SLN+ refers to Positive Sentinel Node
  participants
    N0 | 49
    N1 | 32
    N2 | 12
    N3 | 14
    SLN+ without full axillary dissection | 2
Hormonal Status [Number; unit: participants]
  Estrogen and/or Progesterone Positive | 54
  Estrogen and Progesterone Negative | 55
HER2 Status - Positive [Number; unit: participants] — FISH Amp/IHC refers to fluorescence in situ hybridization amplification/immunohistochemistry
  participants
    FISH Amp/IHC Pos | 93
    FISH Amp/IHC Neg | 8
    FISH Not Amp/IHC Pos | 6
    FISH Not Done/IHC Pos | 2
Left Ventricular Ejection Fraction (LVEF) Measurement [Median (Full Range); unit: percentage] | 63.3 [52 to 78]
Smoking status [Number; unit: participants]
  Never | 60
  Former | 24
  Current | 25
Current use of hypertensive medication [Number; unit: participants]
  Yes | 28
  No | 81
History of diabetes [Number; unit: participants]
  Yes | 10
  No | 99
Menopausal status [Number; unit: participants]
  Premenopausal | 43
  Perimenopausal | 8
  Postmenopausal | 58
Education level [Number; unit: participants]
  Less than high school | 3
  High school | 35
  Beyond high school | 71

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Congestive Heart Failure (CHF) While on Active Treatment
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | AC/PTL
Number analyzed (Participants) | 109
participants | 0

2. Secondary Outcome: Adverse Event Profile as Measured by NCI CTCAE v 3.0
Description: Measured by number of patients with at least one with grade 3+, Grade 4+, Hem, and Non-Hem AEs.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | AC/PTL
Number analyzed (Participants) | 109
Participants
  Grade 3+ Adverse Event | 84
  Grade 4+ Adverse Event | 27
  Grade 3+ Hem Adverse Event | 33
  Grade 4+ Hem Adverse Event | 23
  Grade 3+ Non-Hem Adverse Event | 80
  Grade 4+ Non-Hem Adverse Event | 12

3. Secondary Outcome: Cumulative Incidence (CI) of Cardiac Events
Description: Evaluable patients included those completed the AC phase of their treatment regimen; with post AC cardiac evaluation indicates they are eligible to begin treatment with PTL; and those have begun their post-AC therapy.
  Cardiac events: symptomatic congestive heart failure (CHF), cardiac death and other cardiac events (NCI Common Terminology Criteria for Adverse Events (CTCAE) Grade >=3)
Time Frame: 5 years
Population: 102 patients began post-AC therapy
Measure: Number; unit: Post AC Cardiac Adverse Event
Arm/Group | AC/PTL
Number analyzed (Participants) | 102
Post AC Cardiac Adverse Event | 5

4. Secondary Outcome: Number of Patients Who Experience >= 10 Percent Drop in Left Ventricular Ejection Fraction (LVEF)
Description: Number of Patients Who Experience >= 10 Percent Drop in Left Ventricular Ejection Fraction (LVEF) from baseline to any post-baseline time point.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | AC/PTL
Number analyzed (Participants) | 104
Participants
  Drop ≤ 10 between any 2 time points | 41
  Drop ≥ 10 between any 2 time points | 63

5. Secondary Outcome: Percentage of Participants With Disease-Free Survival (DFS)
Description: DFS was defined as the time from registration to the earliest date of documentation of any local, regional, or distant recurrence of breast cancer (BC); the development of a contralateral BC or second primary other than squamous or basal cell carcinoma of the skin, carcinoma in situ of the cervix, or lobular carcinoma in situ of the breast; or death from any cause without the documentation of one of these events. Participants were followed for a maximum of 5 years from randomization. The median OS with 95%CI was estimated using the Kaplan Meier method.
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AC/PTL
Number analyzed (Participants) | 109
percentage of participants | 91.9 [84.5 to 95.9]

6. Secondary Outcome: Percentage of Participants With Overall Survival (OS)
Description: OS was defined as the time from registration to death of any cause. Participants were followed for a maximum of 5 years from randomization. The median OS with 95%CI was estimated using the Kaplan Meier method.
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AC/PTL
Number analyzed (Participants) | 109
percentage of participants | 95.0 [88.4 to 97.9]

7. Secondary Outcome: Change in Overall LINEAR ANALOGUE SELF ASSESSMENT (LASA) and Change in Symptom Distress Scale (SDS) Overall QOL
Description: LASA score is from 0-90 with 0 being the worst and 90 being the best. SDS score is from 13-65 with 65 being the worst and 13 being the best.
Time Frame: 5 years
Population: Number who completed the QOL questions for each Timeframe.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | AC/PTL
Number analyzed (Participants) | 109
units on a scale
  LASA Time from Cycle 5 Baseline (Months 2-3): number analyzed (Participants) | 102
  LASA Time from Cycle 5 Baseline (Months 2-3) | -11.1 [-14.9 to -7.3]
  LASA Time from Cycle 5 Baseline (Months 5-6): number analyzed (Participants) | 73
  LASA Time from Cycle 5 Baseline (Months 5-6) | -13.2 [-18.2 to -8.1]
  LASA Time from Cycle 5 Baseline (Month 18-Year 3): number analyzed (Participants) | 75
  LASA Time from Cycle 5 Baseline (Month 18-Year 3) | -3.6 [-8.2 to 1.0]
  LASA Time from Cycle 5 Baseline (Year 4-5): number analyzed (Participants) | 57
  LASA Time from Cycle 5 Baseline (Year 4-5) | -0.5 [-5.0 to 4.0]
  SDS Time from Cycle 5 Baseline (Months 2-3): number analyzed (Participants) | 95
  SDS Time from Cycle 5 Baseline (Months 2-3) | -6.7 [-9.2 to -4.3]
  SDS Time from Cycle 5 Baseline (Months 5-6): number analyzed (Participants) | 67
  SDS Time from Cycle 5 Baseline (Months 5-6) | -9.5 [-12.1 to -6.9]
  SDS Time from Cycle 5 Baseline (Month 18-Year 3): number analyzed (Participants) | 70
  SDS Time from Cycle 5 Baseline (Month 18-Year 3) | -1.4 [-4.1 to 1.4]
  SDS Time from Cycle 5 Baseline (Year 4-5): number analyzed (Participants) | 51
  SDS Time from Cycle 5 Baseline (Year 4-5) | 0.3 [-2.5 to 3.1]

8. Secondary Outcome: Proportion of Patients Experienced a Significant Decline in LINEAR ANALOGUE SELF ASSESSMENT (LASA) and a Overall Symptom Distress Scale (SDS) QOL Measurements
Description: Overall Symptom Distress Scale (SDS) QOL Measurement and Overall LINEAR ANALOGUE SELF ASSESSMENT (LASA) QOL Measurement
Time Frame: 5 years
Population: Number who completed the QOL questions for each Timeframe.
Measure: Count of Participants; unit: Participants
Arm/Group | AC/PTL
Number analyzed (Participants) | 109
Participants
  SDS Time from Cycle 5 Baseline (Months 2-3): number analyzed (Participants) | 95
  SDS Time from Cycle 5 Baseline (Months 2-3) | 32
  SDS Time from Cycle 5 Baseline (Months 5-6): number analyzed (Participants) | 67
  SDS Time from Cycle 5 Baseline (Months 5-6) | 33
  SDS Time from Cycle 5 Baseline (Month 18-Year 3): number analyzed (Participants) | 70
  SDS Time from Cycle 5 Baseline (Month 18-Year 3) | 12
  SDS Time from Cycle 5 Baseline (Year 4-5): number analyzed (Participants) | 51
  SDS Time from Cycle 5 Baseline (Year 4-5) | 7
  LASA Time from Cycle 5 Baseline (Months 2-3): number analyzed (Participants) | 102
  LASA Time from Cycle 5 Baseline (Months 2-3) | 67
  LASA Time from Cycle 5 Baseline (Months 5-6): number analyzed (Participants) | 73
  LASA Time from Cycle 5 Baseline (Months 5-6) | 45
  LASA Time from Cycle 5 Baseline (Month 18-3 Year): number analyzed (Participants) | 75
  LASA Time from Cycle 5 Baseline (Month 18-3 Year) | 40
  LASA Time from Cycle 5 Baseline (Year 4-5): number analyzed (Participants) | 57
  LASA Time from Cycle 5 Baseline (Year 4-5) | 19

9. Secondary Outcome: Incidence of Pulmonary Events
Description: Pulmonary events to be included were grade 3 and higher pulmonary adverse events at least possibly related to study treatment, which occur at any time after post-AC treatment is begun, but prior to documentation of a breast cancer recurrence, contralateral breast cancer, secondary primary cancer, non-pulmonary death, or pulmonary death not related to study treatment.
Time Frame: 5 years
Population: No patients experienced grade 3 or higher pulmonary adverse events at least possibly related to study treatment after at any time after post-AC treatment began.
Measure: Number; unit: pulmonary adverse events
Arm/Group | AC/PTL
Number analyzed (Participants) | 109
pulmonary adverse events | 0

ADVERSE EVENTS:
Description: Adverse event data is not available on one patient, thus, only 108 patients were included in adverse events table.
Arm/Group | AC/PTL
Serious Adverse Events (participants affected / at risk) | 17/108
Other Adverse Events (participants affected / at risk) | 107/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AC/PTL (N=108)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (9)
Fatigue (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Leukopenia (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AC/PTL (N=108)
Anemia (Blood and lymphatic system disorders) | 33 (80)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Diastolic dysfunction (Cardiac disorders) | 9 (17)
Left ventricular failure (Cardiac disorders) | 45 (87)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1)
Dry eye (Eye disorders) | 2 (4)
Vision (Eye disorders) | 1 (1)
Vision-Blurred (Eye disorders) | 3 (4)
Watering eyes (Eye disorders) | 1 (3)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Anal hemorrhage (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 93 (426)
Dry mouth (Gastrointestinal disorders) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 9 (16)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 11 (17)
Nausea (Gastrointestinal disorders) | 31 (60)
Oral cavity Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 8 (12)
Oral pain (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 16 (23)
Chills (General disorders) | 2 (2)
Constitutional Symptoms (General disorders) | 1 (1)
Edema limbs (General disorders) | 5 (6)
Fatigue (General disorders) | 101 (624)
Fever (General disorders) | 2 (2)
Influenza Symptoms (General disorders) | 1 (1)
Pain-Chest (General disorders) | 2 (2)
Hypersensitivity (Immune system disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (1)
Dental-tooth infection (Infections and infestations) | 1 (2)
Infection without neutropenia (Infections and infestations) | 3 (5)
Mucosa infection (Infections and infestations) | 1 (2)
Opportunisitic infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sinus infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 3 (4)
Skin (cellulites) infection (Infections and infestations) | 3 (3)
Stomach infection (Infections and infestations) | 1 (1)
Upper airway infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Vaginal infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 2 (3)
Appendix injury (Injury, poisoning and procedural complications) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 20 (60)
Alkaline phosphatase increased (Investigations) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 20 (49)
Leukopenia (Investigations) | 32 (96)
Lymphopenia (Investigations) | 12 (31)
Neutrophil count decreased (Investigations) | 35 (85)
Platelet count decreased (Investigations) | 6 (6)
Weight loss (Investigations) | 4 (15)
Anorexia (Metabolism and nutrition disorders) | 7 (17)
Dehydration (Metabolism and nutrition disorders) | 9 (14)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (5)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 5 (6)
Hyponatremia (Metabolism and nutrition disorders) | 2 (5)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 55 (216)
Bone pain (Musculoskeletal and connective tissue disorders) | 53 (136)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 58 (199)
Dizziness (Nervous system disorders) | 7 (8)
Headache (Nervous system disorders) | 7 (12)
Neuralgia (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 64 (348)
Sinus pain (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Taste (Nervous system disorders) | 6 (16)
Agitation (Psychiatric disorders) | 2 (3)
Anxiety (Psychiatric disorders) | 5 (5)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (6)
Insomnia (Psychiatric disorders) | 6 (9)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1)
Glomerular filtration rate (Renal and urinary disorders) | 1 (1)
Urethra Hemorrhage (Renal and urinary disorders) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 46 (133)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (11)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 53 (177)
Alopecia (Skin and subcutaneous tissue disorders) | 34 (144)
Dermatology (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (6)
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 6 (11)
Nail Changes (Skin and subcutaneous tissue disorders) | 11 (21)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (4)
Sweating (Skin and subcutaneous tissue disorders) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 5 (8)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes